CLINICAL TRIAL: NCT06355037
Title: a Pilot Study to Explore the Efficacy and Safety of Dasatinib Combined With Quercetin to Reverse Chemotherapy Resistance in Triple Negative Breast Cancer.
Brief Title: Dasatinib Combined With Quercetin to Reverse Chemo Resistance in Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024.1.30
Record Dates: First submitted 2024-03-30; First posted 2024-04-09 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Quercetin; Dasatinib; taxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- quercetin and dasatinib (Experimental)
  Interventions: Drug: Quercetin; Drug: Dasatinib; Drug: Taxane/Anthracycline/Eribulin Mesylate/Vinorelbine/Capecitabine/Carboplatin/UTD1/platinum

INTERVENTIONS:
Drug: Quercetin — quercetin 1000mg d1-d3, qw
Drug: Dasatinib — Dasatinib 50mg d1-d3, qw
Drug: Taxane/Anthracycline/Eribulin Mesylate/Vinorelbine/Capecitabine/Carboplatin/UTD1/platinum — Taxane/Anthracycline/Eribulin Mesylate/Vinorelbine/Capecitabine/Carboplatin/UTD1/platinum

SUMMARY:
This is a Phase II, open-label, single-arm study evaluating the efficacy and safety of combined treatment of dasatinib, quercetin with chemotherapy in mTNBC (triple negative breast cancer) patients who progressed during previous chemotherapy.

DETAILED DESCRIPTION:
This is a Phase II, open-label, single-arm study evaluating the efficacy and safety of combined treatment of dasatinib, quercetin with chemotherapy in mTNBC (triple negative breast cancer) patients who progressed during previous chemotherapy. Chemotherapy is the backbone drug for TNBC. How to reverse chemotherapy resistance or how to increase the sensitivity of chemotherapy efficacy, has become an urgent clinical problem to be solved. Our preclinical studies have demonstrated that the combination of dasatinib and quercetin with chemotherapy can effectively eliminate chemotherapy-induced senescent fibroblasts, decrease the proliferation rate of disseminated tumor cells, and ultimately lead to a significant reduction in metastasis and recurrence, thereby enhancing the efficacy of chemotherapy. Based on preclinical studies, the investigators designed this study to enroll mTNBC patients who have progressed during or following chemotherapy, and to explore the efficacy of combined treatment of dasatinib, quercetin with chemotherapy at a clinical level, providing new strategies of combined treatment for TNBC patients.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0, 1
* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
* Radiologic/objective evidence of recurrence or disease progression after chemotherapy for metastatic breast cancer (MBC)
* Adequate hematologic and end-organ function, laboratory test results, obtained within 14 days prior to initiation of study treatment.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures as outlined for each specific treatment arm
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)
* have the cognitive ability to understand the protocol and be willing to participate and to be followed up

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing CNS metastases
* Active or history of autoimmune disease or immune deficiency
* Significant cardiovascular disease
* History of malignancy other than breast cancer within 5 years prior to screening, with the exception of those with a negligible risk of metastasis or death
* Treatment with chemotherapy, radiotherapy,immunotherapy or surgery (outpatient clinic surgery excluded) within 3 weeks prior to initiation of study treatment.
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study
* History of allergies to the drug components of this trial
* Patients who have been using oral steroid hormones for a long time will need to stop for 4 weeks if they have used them occasionally in the past

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Baseline through end of study, assessed up to 6 months
Progression Free Survival (PFS) | Randomization to death from any cause, through the end of study,assessed up to 6 months
Safety and treatment-related AEs | Randomization to death from any cause, through the end of study,assessed up to 12 months
Biomarker analysis1 | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  the pre- and post-treatment levels of age-related secretory factors and neutrophil extracellular traps in serum and lung puncture samples.
Biomarker analysis2 | Baseline until disease progression or loss of clinical benefit, assessed up to 6 months
  Immunohistochemical staining of tissue sections before and after treatment including number of senescent fibroblasts, number and area of neutrophil extracellular traps.

CONTACTS AND LOCATIONS:
Locations (1):
- 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No